CLINICAL TRIAL: NCT00734435
Title: A Proof of Concept, Multi-Center, Randomized, Double-Blind, Parallel, Placebo-Controlled, Study of Zonisamide Sustained Release (SR) 360 mg Versus Placebo in the Prevention of Weight Gain Associated With Olanzapine Therapy for Psychosis
Brief Title: Olanzapine Given in Combination With Zonisamide SR to Prevent Weight Gain in Schizophrenic Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision- Financial Considerations
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OZ-101
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: schizophrenia; schizophreniform; schizoaffective disorder; Zyprexa; olanzapine
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Zonisamide SR 360 mg and olanzapine 10-20 mg daily
  Interventions: Drug: zonisamide SR plus olanzapine
- 2 (Placebo Comparator): Placebo and olanzapine 10-20 mg daily
  Interventions: Drug: Placebo plus olanzapine

INTERVENTIONS:
Drug: zonisamide SR plus olanzapine — zonisamide SR 90 mg given twice daily and olanzapine 10 mg to 20 mg daily for 10 weeks (maintenance period)
  Other Names: Zyprexa
  Arms: 1
Drug: Placebo plus olanzapine — Placebo given twice daily and olanzapine 10-20 mg for 10 weeks (maintenance period)
  Other Names: Zyprexa
  Arms: 2

SUMMARY:
The purpose of this study is to determine if zonisamide SR will prevent weight gain in schizophrenic subjects who take olanzapine (Zyprexa)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects,18-55 years of age
* Outpatients diagnosed with schizophrenia, schizoaffective disorder, or schizophreniform disorder
* Body mass index (BMI) between 22-35 kg/m2 (inclusive)
* Negative serum pregnancy test in women of child-bearing potential
* If women of child-bearing potential, must be non-lactating and agree to use an acceptable form of contraception, which in all cases, includes one type of barrier method, throughout the study period and for 30 days after discontinuation of study drug
* Subject requires a change in antipsychotic treatment and olanzapine is deemed by the Investigator to be a reasonable antipsychotic treatment choice
* No clinically significant abnormality on ECG
* No clinically significant laboratory abnormality
* Negative urine drug screen
* Must be considered reliable and possess a level of understanding that enables the subject to provide written informed consent and to comply with protocol procedures and schedule
* Must be able to read and understand English

Exclusion Criteria:

* Diagnosis of substance dependence within the 6 months prior to randomization
* diagnosis of substance abuse (except for nicotine and caffeine) within the 3 months prior to randomization
* Suicidal behavior or ideation within 3 months prior to randomization, or any current suicidal ideation or intent
* Presence of dementia or other organic brain syndrome
* Serious or unstable medical illnesses
* Known, uncorrected narrow-angle glaucoma
* Diagnosis of eating disorder as defined by DSM-IV within 6 months prior to randomization
* Require treatment with any typical or atypical antipsychotic in addition to olanzapine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Percentage change in total body weight | Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Alan Breier, MD, Principal Investigator — Larue D. Carter Hospital; Mohammed Alam, MD, Principal Investigator — American Medical Research; Gerald Maguire, MD, Principal Investigator — UCI Medical Center; Zinoviy Benzar, MD, Principal Investigator — Brooklyn Medical Institute; Mohammed Bari, MD, Principal Investigator — Synergy Research; Tran Johnson, MD, Principal Investigator — CNRI; Eduard Gfeller, MD, Principal Investigator — Florida Clinical Research Center, Maitland Florida; Andrew Cutler, MD, Principal Investigator — Florida Clinical Research Center, Bradenton Florida; Robert Riesenberg, MD, Principal Investigator — Atlanta Center for Medical Research
Locations (9):
- United States (9):
  - Synergy Research, National City, California
  - UCI Medical Center, Orange, California
  - CNRI San Diego, San Diego, California
  - Florida Clincal Research Center, Bradenton, Florida
  - Florida Clinical Research Center, Maitland, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - American Medical Research, Oak Brook, Illinois
  - Larue D. Carter Hospital, Indianapolis, Indiana
  - Brooklyn Medical Institute, Brooklyn, New York